CLINICAL TRIAL: NCT01575990
Title: Improving Appropriate Colorectal Cancer Screening in Elderly Patients
Brief Title: Elders Preferences in Care Decisions
Acronym: EPIC-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11-1638; P01HS021133-01 (AHRQ)
Record Dates: First submitted 2012-03-29; First posted 2012-04-12 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2015-05

CONDITIONS: Early Detection of Cancer; Colon Cancer; Decision Making; Patient-Centered Care
Keywords: Colon cancer screening; Decision support interventions; Health status; Patient-centered care; Age; Randomized controlled trial; Double blind; UNC
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Making A Decision About CRC Screening (Experimental): A decision support intervention that is a literacy sensitive paper based tool with educational information targeted to the patient's age and gender.
  Interventions: Behavioral: Making A Decision About CRC Screening
- Drivers 65 Plus (Placebo Comparator): The placebo comparator is an attention control with information about driving tips for drivers age 65 and older.
  Interventions: Behavioral: Drivers 65 Plus

INTERVENTIONS:
Behavioral: Making A Decision About CRC Screening — Targeted by age and gender with 3 components.
  1. Educational component
  2. Values clarification exercise
  3. Individualized decision making worksheet
  The intervention or control condition is administered before the index visit with the patient's provider.
  Other Names: Making A Decision About Colon Cancer Screening Woman 70; Making A Decision About Colon Cancer Screening Woman 75; Making A Decision About Colon Cancer Screening Woman 80; Making A Decision About Colon Cancer Screening Men 70; Making A Decision About Colon Cancer Screening Men 75; Making A Decision About Colon Cancer Screening Men 80
  Arms: Making A Decision About CRC Screening
Behavioral: Drivers 65 Plus — This text booklet is provided as an attention control for those in the control arm and like the intervention is administered prior to the index visit with the patient's provider.
  Other Names: Attention control; Control condition
  Arms: Drivers 65 Plus

SUMMARY:
The purpose of this research study is to explore ways to improve appropriate colorectal cancer (CRC) screening in the elderly by attempting to target screening in those most likely to benefit and avoiding screening in those least likely to benefit.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial at the patient level to determine the efficacy of a colorectal cancer screening decision support intervention for patients ages 70 to 84 within a clinical setting. The investigators hypothesize that the use of the intervention will prepare patients for individualized decision making with their providers and result in an improvement in appropriate CRC screening decisions and screening outcomes. To assess appropriate CRC screening decisions and screening, the investigators will use a classification scheme derived from the literature based on age and the Charlson Comorbidity Index. Using this scheme, appropriate screening will include screening for those in the best health because they are likely to benefit, no screening for those in the worst health because they are unlikely to benefit, and evidence of a discussion about CRC screening for those in the intermediate health group because the benefit is unclear.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 70 to 84
* Not up to date with colon cancer screening or surveillance

Exclusion Criteria:

* Men and women younger than 70 years of age or older than 84
* History of Colorectal Cancer
* Inflammatory bowel disease

Ages: 70 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 424 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Appropriate colorectal cancer screening | Six months after intervention or control was adminstered
  The proportion of participants classified as having appropriate colorectal cancer screening in the intervention group compared to the control group. Appropriate screening is a combined outcome measure using patient report of completion or non-completion of CRC screening tests and patient report of discussions about CRC screening with their provider at the index visit. The outcome will be measured six months after the index visit. The index visit is the patient/provider visit that occurred after the decision support intervention or control condition was administered.

SECONDARY OUTCOMES:
Appropriate colorectal cancer screening decisions | At baseline (after intervention or control was administered)
  The proportion of participants classified as having appropriate colorectal cancer screening decisions in the intervention group will be compared to the control group. Appropriate screening decision making is a combined outcome measure using patient report of intent to complete or not complete CRC screening tests and discussions about CRC screening with their provider. This outcome will be measured immediately after the patient and provider index visit. The index visit is the patient/provider visit that occurred after the decision support intervention or control condition was administered.
Appropriate screening and mediators | Six months after intervention or control was adminstered
  For the mediation analysis covariates will be evaluated as potential mediators. The potential mediators to be examined include adequate preparation for individualized decision making (adequate knowledge+ clear values); knowledge scores, screening preference before the index visit, decisional balance, reported discussion during the index visit, gender, previous screening, functional status, and literacy level.
Appropriate screening for health strata | Six months after intervention or control was adminstered
  Once we have tested our hypothesis for the main effects, we will also perform hypothesis-generating exploratory analyses to examine effect of the intervention in sub-groups of patients. We will examine the effect in the three strata (best, intermediate, worst health groups) defined by age and Charlson comorbidity score.
Appropriate screening for stool cards | Six months after intervention or control was adminstered
  For this analysis, appropriate screening test completion will include stool cards for all age groups and health groups. Analyses described for the primary outcome will be performed using this classification of appropriate screening test completion.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Lewis, MD, MPH, Principal Investigator — University of North Carolina; Rowena J Dolor, MD, MHS, Study Director — Duke University
Locations (1):
- Duke Practiced Based Research Network, Durham, North Carolina, United States

REFERENCES:
- [Derived] Dalton AF, Golin CE, Morris C, Kistler CE, Dolor RJ, Bertin KB, Suresh K, Patel SG, Lewis CL. Effect of a Patient Decision Aid on Preferences for Colorectal Cancer Screening Among Older Adults: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244982. doi: 10.1001/jamanetworkopen.2022.44982. PMID 36469317
- [Derived] Lewis CL, Kistler CE, Dalton AF, Morris C, Ferrari R, Barclay C, Brewer NT, Dolor R, Harris R, Vu M, Golin CE. A Decision Aid to Promote Appropriate Colorectal Cancer Screening among Older Adults: A Randomized Controlled Trial. Med Decis Making. 2018 Jul;38(5):614-624. doi: 10.1177/0272989X18773713. PMID 29847251